CLINICAL TRIAL: NCT06088199
Title: A Phase 3, Multi-center, Open-label, Single-arm Study to Assess the Safety of Apremilast (AMG 407) in Pediatric Participants From 6 Through 17 Years of Age With Mild to Moderate Plaque Psoriasis
Brief Title: A Study of Apremilast in Pediatric Participants in Children With Mild to Moderate Plaque Psoriasis
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20200196
Record Dates: First submitted 2023-10-12; First posted 2023-10-18 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-10

CONDITIONS: Plaque Psoriasis
Keywords: Apremilast; Otezla; AMG 407; CC-10004; Pediatric; Plaque psoriasis
MeSH Terms: interventions — apremilast

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Apremilast (Experimental): Apremilast will be dosed by participant's body weight and administered twice daily (BID) in the form of oral tablets, approximately 12 hours apart, without restriction of food or drink.
  Interventions: Drug: Apremilast

INTERVENTIONS:
Drug: Apremilast — Oral tablet
  Other Names: AMG 407; Otezla; CC-10004

SUMMARY:
The primary objective of this post-marketing study is to assess the safety and tolerability of apremilast in pediatric participants (ages 6 through 17 years) with mild to moderate plaque psoriasis.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have a weight of ≥ 20 kg.
* Participant must have an age and sex specific BMI value no lower in range than the fifth percentile on the growth chart for children and adolescents.
* Participant is able to swallow the study medication tablet.
* Diagnosis of chronic plaque psoriasis for at least 6 months prior to screening.
* Has mild to moderate plaque psoriasis at screening and Study Visit 1 as defined by:
* Psoriasis Area Severity Index score 2-15,
* Body surface area 2-15%, and
* Static Physician Global Assessment score of 2-3 (mild to moderate)
* Disease inadequately controlled by or inappropriate for topical therapy for psoriasis.

Exclusion Criteria:

* Guttate, erythrodermic, or pustular psoriasis at screening and Study Day 1.
* Psoriasis flare or rebound within 4 weeks prior to screening.
* Active tuberculosis (TB) or a history of incompletely treated TB per local guidelines.
* History of recurrent significant infections.
* Active infection or infection treated with antibiotic treatment within 14 days of Study Day 1.
* Any history of or active malignancy or myeloproliferative or lymphoproliferative disease.
* Current use of the following therapies that may have a possible effect on psoriasis:
* Conventional systemic therapy for psoriasis within 28 days prior to Study Day 1 (including but not limited to cyclosporine, corticosteroids, methotrexate, oral retinoids, mycophenolate, thioguanine, hydroxyurea, sirolimus, sulfasalazine, azathioprine, and fumaric acid esters).
* Phototherapy treatment (ie, ultraviolet B [UVB], PUVA) within 28 days prior to Study Day 1.
* Biologic therapy:

  * Etanercept (or biosimilar) treatment 28 days prior to Study Day 1
  * Adalimumab (or biosimilar) treatment 10 weeks prior to Study Day 1
  * Other TNF or IL-17 blockers (such as infliximab, certolizumab pegol, secukinumab, ixekizumab, brodalumab, or their biosimilars) within 12 weeks prior to Study Day 1
  * Anti-IL-12 or anti-IL-23 treatment (such as ustekinumab, guselkumab, or tildrakizumab) within 24 weeks prior to Study Day 1.
* Use of tanning booths or other ultraviolet light sources.
* Answer "Yes" to any question on the Columbia-Suicide Severity Rating Scale during screening or at Study Day 1.
* Female participant of childbearing potential with a positive pregnancy test assessed at screening and/or Study Day 1 by a serum and/or urine pregnancy test.

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 51 (Actual)
Dates: Start 2023-10-24 (Actual); Primary Completion 2026-08-06 (Estimated); Study Completion 2026-08-06 (Estimated)

PRIMARY OUTCOMES:
Number of Participants With Treatment-emergent Adverse Events | Day 1 up to approximately 285 days

SECONDARY OUTCOMES:
Growth and Development as Assessed by Height | Day 1 up to approximately 285 days
Growth and Development as Assessed by Weight | Day 1 up to approximately 285 days
Growth and Development as Assessed by Body Mass Index (BMI) | Day 1 up to approximately 285 days
Columbia-Suicide Severity rating Scale (C-SSRS) | Day 1 to Day 225
Tanner Staging of Sexual Maturity | Day 1 and Day 225
Number of Participants With Psoriasis Flare | Up to approximately 285 days
Number of Participants With Psoriasis Rebound | Up to approximately 285 days
Number of Participants Experiencing Diarrhea Sympotms as Assessed by Stool Diaries | Day 1 to Day 225
Number of Participants with Clinically Significant Changes in Laboratory Parameters | Up to approximately 225 days
Number of Participants with Clinically Significant Changes in Vital Signs | Up to approximately 285 days

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (30):
- United States (30):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Affiliated Dermatology, Scottsdale, Arizona
  - Clear Dermatology, Scottsdale, Arizona
  - Johnson Dermatology Clinic, Fort Smith, Arkansas
  - Avance Clinical Trials, Laguna Niguel, California
  - University of California Irvine, Orange, California
  - MedDerm Associates, San Diego, California
  - Clinical Science Institute, Santa Monica, California
  - California Dermatology Institute, Thousand Oaks, California
  - Pediatric Skin Research LLC, Coral Gables, Florida
  - Ciocca Dermatology, Miami, Florida
  - University of South Florida, Tampa, Florida
  - Endeavor Health Clinical Trials Center, Skokie, Illinois
  - Dawes Fretzin Clinical Research Group, LLC, Indianapolis, Indiana
  - Southern Indiana Clinical Trials, New Albany, Indiana
  - Great Lakes Research Group Inc- Sheffield, Bay City, Michigan
  - Henry Ford Medical Center - New Center One, Detroit, Michigan
  - Dermatology and Skin Cancer Center of Lees Summit, Lee's Summit, Missouri
  - Boeson Research, Missoula, Montana
  - Empire Dermatology, East Syracuse, New York
  - State University of New York, Downstate Medical Center, Manhasset, New York
  - OptiSkin Medical, New York, New York
  - Hightower Clinical LLC, Oklahoma City, Oklahoma
  - Dermatology Research Center of Oklahoma, PLLC, Tulsa, Oklahoma
  - Oregon Health and Science University, Portland, Oregon
  - Medical University of South Carolina, Charleston, South Carolina
  - Studies in Dermatology LLC, Cypress, Texas
  - Austin Institute for Clinical Research, Pflugerville, Texas
  - Stride Clinical Research LLC, Sugar Land, Texas
  - Frontier Derm Partners, Mill Creek, Washington

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors. If not approved, a Data Sharing Independent Review Panel will arbitrate and make the final decision. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: http://www.amgen.com/datasharing

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com